CLINICAL TRIAL: NCT06761352
Title: Questionnaire About Risk Factors of Iron Deficiency Anemia in Pregnancy and How to Prevent it
Brief Title: Questionnaire About Risk Factors of Iron Deficiency Anemia in Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Sayed Hussien, Invstigator doctor, Assiut University
Other Study IDs: Iron deficiency anemia in preg
Record Dates: First submitted 2024-12-24; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Iron Deficiency Anaemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anemia in pregnancy,and especially iron deficiency anemia is both a long standing scholarly interest ,the aim of my research to summarise the risk factors of iron deficiency anemia in pregnancy, especially in Egypt as a less developed country,and suggest recommendations about how to prevent it

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older with established iron deficiency anemia (HB less than 10)
* established intrauterine pregnancy
* women want to participate in the study

Exclusion Criteria:

* anemia due to other causes
* recent blood transfusion in the last 3 months
* women with threatened miscarriage
* women are known to have pathological blood loss (urinary bleeding or GIT bleeding) 5- history of haematological disorder 6- women used iron in the past 3 months

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women attending Assiut university hospital for antenatal care
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Risk factors of iron deficiency anemia in pregnancy | 1 Year